CLINICAL TRIAL: NCT00685464
Title: Intravenous vs. Intracoronary Use of Abciximab
Brief Title: Intravenous Versus Intracoronary Use of Abciximab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Jan Skov Jensen, MD, Ph.D, DMSc, Gentofte University Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: UHGentofte
Record Dates: First submitted 2008-05-22; First posted 2008-05-28 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2009-02

CONDITIONS: Atherosclerosis; Ischemic Heart Disease
Keywords: Abciximab; Reo-Pro; Intracoronary; PCI
MeSH Terms: conditions — Atherosclerosis; Myocardial Ischemia | interventions — Abciximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator): Intravenous bolus Abciximab.
  Interventions: Drug: Abciximab
- Abciximab (Active Comparator): Intracoronary bolus abciximab.
  Interventions: Drug: Abciximab

INTERVENTIONS:
Drug: Abciximab — Intravenous.
  Arms: 2
Drug: Abciximab — Intracoronary
  Arms: Abciximab

SUMMARY:
The aim of this study is to investigate wether intracoronary use of bolus Abciximab is superior to intravenous bolus in patients undergoing percutaneous coronary intervention.

DETAILED DESCRIPTION:
STEMI patients with indication for adjuvant therapy with GPI during pPCI, and who gave informed consent, were randomized, using sealed, opaque envelopes, to either IC or IV bolus (0.25 mg/kg body weight) followed by a 12-hour IV infusion of abciximab (0.125 μg/kg body weight per minute). IC bolus of abciximab was delivered via the PCI guiding catheter directly into the culprit artery, whereas IV bolus was given in a peripheral vein, both after filtering of the drug. The drug of use in our centre is Reo-Pro® manufactured by Eli Lilly, Denmark, who had no involvement, economically or scientifically, in the trial.

Inclusion criteria in the present analysis were STEMI (onset of chest pain ≤ 12 hours and ST-segment elevation in two contiguous leads of ≥ 2 mm in V1-V3 or ≥ 1 mm in other leads), age ≥ 18 years and indication for adjuvant therapy with abciximab (e.g. as bail-out in case of no-reflow, high thrombus burden, dissection, or type B2/C lesions) on the operator's discretion.

Exclusion criteria were known allergy to abciximab, ongoing bleeding, recent stroke, major surgery within 2 months, known bleeding disorder, or pregnancy.

All patients were pre-treated with oral Aspirin (300-500 mg) and Clopidogrel (300-600 mg) and 10,000 IU of unfractionated heparin given IV as a single-dose according to national guidelines for STEMI patients referred for pPCI. Patients were discharged with life-long Aspirin in a dose of 75 mg/day and Clopidogrel for 12 months in a dose of 75 mg/day.

In relation to PCI the following data were recorded: infarct localization on ECG and coronary angiography, number of diseased vessels, TIMI flow before and after PCI, lesion type (A, B, C), and type and number of stents implanted.

Furthermore, the following baseline data were registered: age, gender, hypertension (defined as being treated with blood pressure lowering medication, or being diagnosed as having hypertension during hospital stay, i.e. systolic blood pressure > 140 mmHg, or diastolic blood pressure > 90 mmHg), hypercholesterolemia (defined as being treated with lipid lowering medication, or having an in-hospital fasting total cholesterol of ≥ 5 mmol/L (192 mg/dL), or LDL ≥ 3 mmol/L (116 mg/dL)), smoking status, family history of coronary heart disease, diabetes (defined as being treated with an anti-diabetic agent, or having an in-hospital fasting plasma glucose ≥ 6.1 mmol/L, or a non-fasting plasma glucose ≥ 11.1 mmol/L), prior coronary vessel disease, and height and weight. Medication status was recorded at admission, at discharge, and at the 30-day follow up. Left ventricular ejection fraction (LVEF) was assessed during hospital stay by echocardiography using the 16 standard segments model (28).

Primary end-points were defined as death and target vessel revascularization (TVR).

Furthermore recurrent myocardial infarction (MI) and stroke within the first 30 days were recorded. Bleeding complications were recorded during hospital stay. Minor bleeding complications were defined as bleedings from the vascular access site, not requiring blood transfusion, but leading to premature (< 12 hours) cessation of the abciximab IV infusion.

Major bleeding complications were defined as bleedings that required cessation of abciximab infusion and subsequent blood transfusion and/or vascular surgery.

After 30 days patients were contacted by telephone, subsidiary by letter. All possible events within this period were confirmed by checking hospital source data. All end-points were evaluated by an independent committee that was unaware of study-group assignment. No patients were lost to follow up.

All patients gave written informed consent. The study was approved by the local ethics committee and the Danish Medicines Agency and carried out in concordance with the Helsinki-II Declaration and the GCP requirements.

ELIGIBILITY:
Inclusion Criteria:

* Usually inclusion criteria for Abciximab, that is:
* Adjunct to PCI for the prevention of cardiac ischemic complications:

  * In patients undergoing PCI
  * In patients with UA not responding to conventional medical therapy when PCI is planned within 24 hours

Exclusion Criteria:

Usually exclusion criteria for Abciximab, that is:

* Active internal bleeding, recent (within 6 weeks) gastrointestinal (GI) or genitourinary (GU) bleeding of clinical significance
* History of cerebrovascular accident (CVA) within 2 years, or CVA with a significant residual neurological deficit
* Bleeding diathesis
* Administration of oral anticoagulants within 7 days unless prothrombin time is less than or equal to 1.2 times control, thrombocytopenia (<100,000 cells/µL)
* Recent (within 6 weeks) major surgery or trauma
* Intracranial neoplasm
* Arteriovenous malformation, or aneurysm
* Severe uncontrolled hypertension
* Presumed or documented history of vasculitis
* Use of intravenous dextran before percutaneous coronary intervention, or intent to use it during intervention
* Known hypersensitivity to any component of this product or to murine proteins.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2006-01; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Death, TVR, bleeding, stroke | 30 days and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Allan Iversen, MD, Principal Investigator — Gentofte University Hospital
Locations (1):
- Dept. of Cardiology, Gentofte University Hospital, Hellerup, Denmark